CLINICAL TRIAL: NCT01865305
Title: A Randomised, Double-blind, Multiple Period Crossover Trial Comparing Insulin 454 and Insulin Aspart Premixes With Separately Injected, Simultaneous Doses of Insulin 454 and Insulin Aspart, Compared With Biphasic Insulin Aspart 30 (NovoMix® 30) in Male Subjects With Type 1 and Type 2 Diabetes Mellitus
Brief Title: Comparison of Explorative Formulation of Insulin Degludec and Insulin Aspart Co-formulation Versus Explorative Formulation of Insulin Degludec and Insulin Aspart Separately Compared With Biphasic Insulin Aspart 30 in Male Subjects With Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN5401-1738; 2006-002430-37 (EudraCT Number)
Record Dates: First submitted 2013-05-27; First posted 2013-05-30 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — insulin degludec; Insulin Aspart; insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trial part 1 (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart 30; Drug: insulin degludec/insulin aspart 40; Drug: insulin degludec/insulin aspart 50; Drug: insulin degludec; Drug: insulin aspart; Drug: biphasic insulin aspart 30
- Trial part 2 (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart 40; Drug: insulin degludec/insulin aspart 50; Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: insulin degludec/insulin aspart 30 — Single dose administrated subcutaneously (s.c., under the skin).
  Arms: Trial part 1
Drug: insulin degludec/insulin aspart 40 — Single dose administrated subcutaneously (s.c., under the skin).
  Arms: Trial part 1
Drug: insulin degludec/insulin aspart 50 — Single dose administrated subcutaneously (s.c., under the skin).
  Arms: Trial part 1
Drug: insulin degludec — Single dose administrated subcutaneously (s.c., under the skin).
  Arms: Trial part 1
Drug: insulin aspart — Single dose administrated subcutaneously (s.c., under the skin).
  Arms: Trial part 1
Drug: biphasic insulin aspart 30 — Single dose administrated subcutaneously (s.c., under the skin) as comparator.
  Arms: Trial part 1
Drug: insulin degludec/insulin aspart 40 — Single dose administrated subcutaneously (s.c., under the skin).
  Arms: Trial part 2
Drug: insulin degludec/insulin aspart 50 — Single dose administrated subcutaneously (s.c., under the skin).
  Arms: Trial part 2
Drug: biphasic insulin aspart 30 — Single dose administrated subcutaneously (s.c., under the skin).
  Arms: Trial part 2

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to compare different ratios of explorative formulations, not similar to the proposed commercial formulation, of IDegAsp (co-formulation of insulin degludec/insulin aspart and insulin aspart) with separately injected, simultaneous doses of insulin degludec (insulin 454), and insulin aspart, compared with biphasic insulin aspart 30 in male subjects with type 1 and type 2 diabetes mellitus.

Trial part 1 is a five-period cross-over trial with incomplete block-design in subjects with type 1 diabetes where each subject will be randomised to five out of the ten possible treatments. Each treatment consists of an injection of the insulin product followed by a euglycemic clamp with a washout period of 7-15 days between treatments.

Trial part 2 is a three-period cross-over trial with complete blockdesign in subjects with type 2 diabetes. Each treatment consists of an injection of the insulin product followed by a euglycaemic clamp with a washout period of 7-15 days between treatments.

ELIGIBILITY:
Inclusion Criteria:

* The subject will be a male volunteer, who is considered to be generally healthy, except for underlying diabetes mellitus and concomitant medical complications (e.g. hypertension) based on an assessment of medical history, physical examination and clinical laboratory data, as judged by the Investigator
* Glycosylated haemoglobin A1c (HbA1c) below or equal to 10 % based on central laboratory results
* ADDITIONAL INCLUSION CRITERA FOR SUBJECTS WITH TYPE 1 DIABETES:
* Diagnosed with type 1 diabetes mellitus and treated with insulin for at least 12 months
* Body Mass Index (BMI) between 18.0 and 27.0 kg/m^2 (both inclusive)
* ADDITIONAL INCLUSION CRITERA FOR SUBJECTS WITH TYPE 2 DIABETES:
* Diagnosed with type 2 diabetes mellitus for at least 12 months
* Treated with insulin for the last 3 months prior to screening.
* Body Mass Index (BMI) between 22.0 and 35.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* A subject with a history of significant multiple drug allergies or with a known or suspected allergy to the trial product or any medicine chemically related to the trial product, as judged by the Investigator
* A subject who has participated in any other trials involving investigational products within the 3 months preceding the start of dosing

Ages: 18 Years to 69 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2006-09; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Area under the insulin aspart concentration curve from 0-2 hours (for subjects with type 1 diabetes) | 0-2 hours after dosing
Maximum glucose infusion rate divided by the average glucose infusion rate (for subjects with type 2 diabetes) | 0-24 hours after dosing

SECONDARY OUTCOMES:
Area under the glucose infusion rate curve | 0-24 hours after dosing
Area under the serum insulin degludec concentration curve | 0-96 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com